CLINICAL TRIAL: NCT03767153
Title: Clinical Evaluation of the Safety and Performance of Fractional Radiofrequency for the Treatment and Reduction of Acne Scarring
Brief Title: Clinical Evaluation of Fractional Radiofrequency for the Treatment of Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VI1018
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Acne Scars
Keywords: acne scarring; acne scar; fractional radiofrequency; fractional RF

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of photographs taken at baseline and 6, 12 weeks post final treatment by independent evaluators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 80 pin applicator (Experimental)
  Interventions: Device: Venus Viva
- 160 pin applicator (Active Comparator)
  Interventions: Device: Venus Viva

INTERVENTIONS:
Device: Venus Viva — The Venus Viva™ fractional RF applicator has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars.
  Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart. The left and right side of the face will be treated and assessed as independent sites, and the same applicator tip configuration will be used to treat both sides at all 3 treatment visits.

SUMMARY:
Prospective, single centre, evaluator-blind study of the safety and performance of fractional radiofrequency (RF) for the treatment and reduction of acne scarring. The study will evaluate 50 treatment sites in subjects requesting treatment of their acne scarring. The study will involve three treatments on both sides of the face with 3-5 week intervals between each treatment. Subjects will be followed at 6 and 12 weeks after their last treatment. Analysis will be performed on all subjects who receive at least one treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects 22 years of age or over who are seeking treatment and reduction of their facial acne scarring.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Implantable defibrillators, cardiac pacemakers, and other metal implants
2. Subjects with any implantable metal device in the treatment area
3. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
4. Permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
5. Current or history of any kind of cancer, or pre-malignant moles.
6. Severe concurrent conditions, such as cardiac disorders.
7. Pregnancy or intending to become pregnant during the study and nursing.
8. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
9. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only after a prophylactic regime has been followed for 2 weeks or longer prior to enrollment, or according to Investigator's discretion .
10. Poorly controlled endocrine disorders, such as diabetes.
11. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
12. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
13. History of bleeding coagulopathies, or use of anticoagulants (excluding daily aspirin).
14. Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last three months, if face is treated.
15. Use of isotretinoin (Accutane®) or other retinoids within six months prior to treatment or as per physician's discretion.
16. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g. ibuprofen-containing agents) one week before and after each treatment session.
17. Any surgical procedure in the treatment area within the last six months or before complete healing.
18. Treating over tattoo or permanent makeup.
19. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.
20. As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, Study Director — Venus Concept
Locations (1):
- Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Port Orange, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 Pin Applicator | 160 Pin Applicator | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.5) | 45.0 (10.1) | 45.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 9 | 19
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Acne Scar Improvement Assessed by the Global Aesthetic Improvement Scale (GAIS) at 12 Weeks.
Description: Evaluate the efficacy of overall facial acne scar improvement assessed live by the Investigator and a subject assessment of facial appearance including the Global Aesthetic Improvement Scale (GAIS).
  The Global Aesthetic Improvement Scale is a seven-grade subjective test.
  Three independent evaluators evaluated before and after photographs and graded them for change.
  Possible responses were (3) Very Much Improved, (2) Much Improved, (1) Improved, (0) No Change, (-1) Worse, (-2) Much Worse, and (-3) Very Much Worse. For reporting of outcomes, the higher the GAIS value, the greater the improvement (Range -3 to 3).
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
Number analyzed (Participants) | 14 | 11
score on a scale | 1.06 (0.13) | 0.85 (0.13)

2. Secondary Outcome: Subject Satisfaction
Description: Subjects' assessment of satisfaction with the treatment using a 5 point Subject Satisfaction Scale at 6 Weeks and 12 weeks post-treatment.
  The Subject Satisfaction Scale is a five-grade subjective test.
  Participant were asked their satisfaction level post treatment.
  Possible responses were (4) Very Satisfied, (3) Satisfied, (2) Having No Opinion, (1) Unsatisfied, and (0) Very Unsatisfied.
Time Frame: 6 Weeks and 12 Weeks Post- Final Treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
Number analyzed (Participants) | 14 | 11
score on a scale
  6-weeks | 3.25 (0.18) | 3.55 (0.21)
  12-weeks | 3.18 (0.18) | 3.36 (0.24)

3. Secondary Outcome: Subject Scale - Visual Analog Scale for Pain
Description: Subject's assessment of discomfort and pain after treatments as measured by a 10 cm visual analog scale (VAS).
  The Visual Analog Scale is a scale from 0 cm (no pain) and 10 cm (pain as bad as it can be).
  Possible responses were of 0 to 0.4 cm can be considered (no pain); 0.5 to 4.4 cm (mild pain), 4.5 to 7.4 cm (moderate pain), and 7.5 to 10 cm (severe pain).
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Error); unit: cm
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
Number analyzed (Participants) | 14 | 11
cm | 2.23 (0.26) | 2.05 (0.27)

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events [Safety]
Description: Subjects experiencing a treatment-related adverse event (AE) by 12 weeks post-treatment.
Time Frame: Up to 12 Weeks Post-Final Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
Number analyzed (Participants) | 14 | 11
Participants | 0 | 0

5. Secondary Outcome: Subject Scale - 5 Point Scale for Treatment Tolerability
Description: Subject's assessment of treatment tolerability as measured by a 5 point scale.
  Participant were asked their tolerability level post treatment.
  Possible scores were; (4) Very Tolerable, (3) Tolerable, (2) Having No Opinion, (1) Intolerable, and (0) Very Intolerable.
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
Number analyzed (Participants) | 14 | 11
score on a scale | 3.36 (0.07) | 3.48 (0.06)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | 80 Pin Applicator | 160 Pin Applicator
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT03767153/Prot_SAP_000.pdf